CLINICAL TRIAL: NCT01008865
Title: A Randomized Comparison of the Studer Pouch vs. the T-Pouch Orthotopic Neobladder Urinary Diversion in Bladder Cancer Patients
Brief Title: A Comparison of the Studer Pouch Versus the T-Pouch Orthotopic Neobladder Urinary Diversion in Bladder Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4B-01-2
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Studer Pouch (Experimental): Studer Pouch orthotopic urinary diversion
  Interventions: Procedure: Studer Pouch orthotopic urinary diversion
- T-Pouch (Experimental): T-Pouch orthotopic urinary diversion
  Interventions: Procedure: T-Pouch orthotopic urinary diversion

INTERVENTIONS:
Procedure: Studer Pouch orthotopic urinary diversion
  Arms: Studer Pouch
Procedure: T-Pouch orthotopic urinary diversion
  Arms: T-Pouch

SUMMARY:
This is a prospective, randomized study of two types of continent ileal neobladder construction in patients undergoing cystectomy for primary bladder cancer. Patients will be randomly assigned to have either a T-pouch or a Studer pouch constructed at the time of their surgery. They will be followed long-term to determine the relative advantages and disadvantages of the two types of diversion. The investigators' hypothesis is that the inclusion of an antireflux mechanism in the T-pouch will result in significantly fewer episodes of symptomatic urinary tract infection, and will have a lower incidence of upper tract dilation and loss of renal function over the long term.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing radical cystectomy for bladder cancer who are considered candidates for a neobladder reconstruction are eligible for enrollment.
* Diagnosed with primary bladder cancer (any histology).
* Scheduled to undergo a radical cystectomy (cystoprostatectomy in men and anterior exenteration in women).
* Felt by the treating physician to be a candidate for an orthotopic neobladder urinary diversion.
* Be competent and willing to sign the informed consent.
* Patients may have received previous radiation therapy or intravesical or systemic chemotherapy. Patients with documented metastatic disease are not excluded as long as they are felt to be candidates for a continent neobladder urinary diversion.

Exclusion Criteria:

* Patients undergoing radical cystectomy for any malignancy other than primary bladder cancer (for example prostate cancer or colon cancer invading the bladder,or a gynecologic malignancy), or non-malignant disease (such as a neurogenic bladder or radiation cystitis).
* Unwilling or unable to sign the informed consent.
* Not eligible for an orthotopic neobladder reconstruction.
* A history of other malignancy (except for stage I cancer treated with curative intent without evidence of recurrence, clinically localized prostate cancer either untreated or treated with prostatectomy or radiation therapy or hormone therapy,or non-melanoma skin cancer) within the previous 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2002-01-04 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the long-term outcome (> 3 years) as it pertains to renal function, anatomy of the upper urinary tracts, and the requirement for medical or surgical intervention (ie for symptomatic urinary tract infections). | 3 years after date of last patient enrolled

SECONDARY OUTCOMES:
A secondary endpoint is the length of surgery and the incidence of early postoperative complications (<30 days from surgery) believed to be related to the type of urinary diversion. | Within 30 days after surgery
An additional secondary endpoint is cancer recurrence and overall survival, which will be recorded in each patient. | Yearly for the first 5 years, then every 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Daneshmand, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States